CLINICAL TRIAL: NCT05106738
Title: Phase Angle as a New Possible Prognostic Factor in Chronic Intestinal Inflammatory Diseases
Brief Title: Phase Angle and Chronic Intestinal Inflammatory Diseases
Acronym: PHIBO
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Associate Professor, University of Bari
Other Study IDs: Policlinic hospital, 9
Record Dates: First submitted 2021-10-23; First posted 2021-11-04 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Diseases; Mucosal Inflammation; Leukocyte L1 Antigen Complex; C-Reactive Protein
MeSH Terms: conditions — Inflammatory Bowel Diseases; Mucositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phase angle (PhA) is a biometric parameter measured by bioimpedance analysis (BIA), which reflects organism cellularity and tissues hydration. In addition, since it correlates with the presence of inflammation and the nutritional status, it could be useful to monitor inflammatory bowel disease (IBD) activity. The aim of this study was to establish the potential use of PhA as a new non-invasive and sensitive marker correlated with mucosal healing and/or IBD activity.

DETAILED DESCRIPTION:
Currently, fecal calprotectin is considered the best indirect marker inversely correlated with the mucosal healing in patients with inflammatory bowel disease (IBD). C reactive protein (CRP), is less reliable than fecal calprotectin in the evaluation of IBD activity. In order to establish the potential use of phase angle (PhA) as a new non-invasive and sensitive marker of mucosal healing and/or disease activity in patients with IBD, patients with diagnosis of chronic inflammatory bowel diseases (IBD) according to the European Crohn's and Colitis Organization (ECCO) guidelines will be enrolled. In these patients, the following parameters will be evaluated: age, sex, body mass index (BMI), percentage of weight loss in the last 6 months, duration of illness, location of disease, any previous intestinal surgery, ongoing therapy for IBD, activity disease by clinical scores, CRP, fecal calprotectin, disease activity by endoscopic scores, PhA and fat free mass (FFM).

ELIGIBILITY:
Inclusion Criteria:

* histological report confirming the diagnosis of IBD,
* value of C-reactive protein (CRP)
* fecal calprotectin,
* colonoscopy within 3 months from the enrollment.

Exclusion Criteria:

* presence of ascites or edema,
* chronic or autoimmune inflammatory diseases,
* ongoing infections,
* recent surgery (in the last 6 months),
* neoplastic diseases,
* ongoing enteral or parenteral nutrition,
* presence of fistulae,
* ileostomy or colostomy,
* short bowel syndrome,
* pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease and patients with Ulcerative Colitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The correlation of phase angle with mucosal healing in patients with inflammatory bowel disease | At enrollment
  The evaluation of phase angle (PhA), expressed in degrees, will be obtained by bioimpedenziometry, using a specific software (Bodygram Pro 3.0, Akern srl, Pontassieve, Italy). The assessment of mucosal healing will be performed by the following endoscopic scores: the Simple Endoscopic Score for Crohn's Disease (SES-CD) and the Mayo endoscopic score for Crohn's disease and Ulcerative Colitis (UC), respectively.

SECONDARY OUTCOMES:
Evaluation of the presence of malnutrition by bioimpedance analysis | At enrollment
  Malnutrition will be assessed by the evaluation of body composition [fat free mass (FFM) and fat mass (FM) expressed in kg], by bioimpedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michele Barone, MD, Principal Investigator — University of Bari
Locations (1):
- Michele Barone, Bari, BA, Italy